CLINICAL TRIAL: NCT03564106
Title: Comparison Between Intra-articular Pulsed Radiofrequency With Steroids Injection Versus Intra-articular Steroids Injection in Chronic Sacroiliac Joint Arthritis
Brief Title: Intra-articular Pulsed Radiofrequency With Steroids Injection Versus Intra-articular Steroids Injection in Chronic Sacroiliac Joint Arthritis
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ghada Mohammed AboelFadl, Principal Investigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 17200203
Record Dates: First submitted 2018-06-02; First posted 2018-06-20 (Actual); Last update posted 2021-01-20 (Actual); Status verified 2021-01

CONDITIONS: Pain Management
Keywords: chronic sacroilitis,radiofrequancy,intraarticular steroids injection
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group A (Experimental): receive intraarticular radiofrequency + methylprednisolone (30 mg)
  Interventions: Drug: intraarticular radiofrequency + intraarticular methylprednisolone
- group C (Experimental): receive intraarticular methylprednisolone (30 mg)
  Interventions: Drug: intraarticular methylprednisolone

INTERVENTIONS:
Drug: intraarticular radiofrequency + intraarticular methylprednisolone — intraarticular radiofrequency + intraarticular methylprednisolone (30 mg)
  Arms: group A
Drug: intraarticular methylprednisolone — intraarticular methylprednisolone (30 mg)
  Arms: group C

SUMMARY:
The sacroiliac joint is Located between the pelvis and base of the spine, the sacroiliac joints are strong, stable joints that allow for little movement. While these joints do not bend like a knuckle or knee, they are susceptible to degenerative arthritis. Sacroiliac joint pain is one of the most common causes of chronic low back pain, accounting for 10% to 27% of patients with chronic lower back pain. It is known to be caused by abnormal motion in this joint, namely, too much motion or too little motion. Patients with pain experience various degrees of pain in the low back, groin, buttock, or posterior thigh.

DETAILED DESCRIPTION:
The pain starts when the Sacroiliac joint gets inflamed. There are several reasons it could happen. It could be hurt when playing sports or if fall down.

Sometimes start hurting when the ligaments that hold the SI joint together are damaged, which may make the joint move abnormally. The pain associated with sacroiliitis most commonly occurs in the buttocks and lower back. It can also affect the legs, groin and even the feet.

ELIGIBILITY:
Inclusion Criteria:

* All patients must have chronic pain more than 6 months and have failed medical treatment.

Exclusion Criteria:

* Infection at the site of injection
* Opioids addiction
* Coagulopathy or another bleeding diathesis
* Those who refuse to participate in the study
* Ankylosing Spondylitis patients

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2021-01-01 (Actual); Study Completion 2021-01-15 (Actual)

PRIMARY OUTCOMES:
pain intensity | up to 6 months
  Numeric Rating Scale (NRS)

SECONDARY OUTCOMES:
Patient Impression | up to 6 months
  Patient Global Impression of Change Scale (PGIC)
Pain Disability | up to 6 months
  Pain Disability Index ( PDI)

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut governorate, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bogduk N. Pulsed radiofrequency. Pain Med. 2006 Sep-Oct;7(5):396-407. doi: 10.1111/j.1526-4637.2006.00210.x. No abstract available. PMID 17014598
- [Background] Borowsky CD, Fagen G. Sources of sacroiliac region pain: insights gained from a study comparing standard intra-articular injection with a technique combining intra- and peri-articular injection. Arch Phys Med Rehabil. 2008 Nov;89(11):2048-56. doi: 10.1016/j.apmr.2008.06.006. PMID 18996232
- [Background] Choi WJ, Hwang SJ, Song JG, Leem JG, Kang YU, Park PH, Shin JW. Radiofrequency treatment relieves chronic knee osteoarthritis pain: a double-blind randomized controlled trial. Pain. 2011 Mar;152(3):481-487. doi: 10.1016/j.pain.2010.09.029. Epub 2010 Nov 4. PMID 21055873
- [Background] Do KH, Ahn SH, Jones R, Jang SH, Son SM, Lee DG, Cho HK, Choi GS, Cho YW. A New Sacroiliac Joint Injection Technique and Its Short-Term Effect on Chronic Sacroiliac Region Pain. Pain Med. 2016 Oct;17(10):1809-1813. doi: 10.1093/pm/pnw003. Epub 2016 Feb 25. PMID 27738191